CLINICAL TRIAL: NCT01318278
Title: Dopamine Versus Vasopressin for Cardiovascular Support in Extremely Low Birth Weight Infants: A Randomized, Blinded Pilot Study
Brief Title: Study of Dopamine Versus Vasopressin for Treatment of Low Blood Pressure in Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Danielle Rios, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-27661
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Hypotension
Keywords: Hypotension; Low blood pressure; Neonate; Dopamine; Vasopressin; Extremely Low Birth Weight Infant
MeSH Terms: conditions — Hypotension; Diabetes Insipidus | interventions — Dopamine; Arginine Vasopressin; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dopamine treatment (Active Comparator): Dopamine treatment beginning at 5 mcg/kg/min and titrated by 5 mcg/kg/min to effect up to maximum of 20 mcg/kg/min
  Interventions: Drug: Dopamine
- Vasopressin treatment (Active Comparator): Arginine Vasopressin treatment beginning at 0.01 units/kg/hr and titrated up by 0.01 units/kg/hr to effect up to a maximum of 0.04 units/kg/hr
  Interventions: Drug: Arginine Vasopressin
- Comparison Arm (No Intervention): Infants who did not require vasopressor support for hypotension during the first 24 hours of life

INTERVENTIONS:
Drug: Dopamine — dopamine at low/medium/and high dose (5, 10, 15, and 20 mcg/kg/min) given IV as a continuous infusion, titrated up for efficacy
  Other Names: Dopamine Hydrochloride
  Arms: Dopamine treatment
Drug: Arginine Vasopressin — vasopressin at low/medium/and high dose (0.01, 0.02, 0.03, or 0.04 units/kg/hr) given IV as a continuous infusion, titrated up for efficacy
  Other Names: Vasopressin; Antidiuretic Hormone (ADH); Pitressin (US brand name); Pressyn;Pressyn AR (Canadian brand names); Argipressin
  Arms: Vasopressin treatment

SUMMARY:
Low blood pressure or hypotension is a very important problem that is often seen in premature babies, especially those with low birth weight. Severe hypotension leads to significant problems including brain bleeds, developmental delays, kidney and liver problems, and other issues that can affect babies for the rest of their lives. An important aspect in the management of infants with hypotension is the decision of when to treat and with what agent. Research is being conducted to try to find the best medication to use in these situations. Dopamine is often used first, but it does not always prove to be effective, and it has several concerning side effects. This study will look at vasopressin, which has fewer side effects, as a first-line medication for low blood pressure in extremely low birth weight infants.

Hypotheses and Specific Aims: This study will show superiority of vasopressin to dopamine in preterm, extremely low birth weight infants who have hypotension within the first 24 hours of life. We will specifically look at its ability to raise blood pressure values, improve clinical symptoms seen, any adverse effects, and clinical outcomes of babies being treated.

DETAILED DESCRIPTION:
Hypotension in the low birth weight (LBW) and extremely low birth weight (ELBW) infant is often encountered in the postnatal adaptation phase. Severe, prolonged hypotension contributes to cellular dysfunction and cell death. Systemic hypotension affects close to half of all ELBW infants and a significant portion of LBW infants. The true definition of hypotension remains to be a question. There is a linear association between birth weight, gestational age, and mean blood pressure but blood pressure can vary significantly in the first day of life. The critical period tends to be the first 24-36 hours of life as blood pressure tends to rise significantly in the first 72 hours of life regardless of gestational age. Preterm infants suffering from hypotension have a higher incidence and increased severity of intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), and long-term neurodevelopmental sequelae compared to normotensive preterm infants. Effects on other organ systems can result in renal injury, hepatic injury, and the development of necrotizing enterocolitis among other complications. An important aspect in the management of infants with hypotension is the decision of when to treat and with what agent. Dopamine is commonly used as first-line therapy, but issues with efficacy and its side effect profile have lessened its favorability over the years. Few studies compare dopamine to other agents as a first -line treatment. This study hopes to contribute to the literature information on vasopressin as a potential first-line agent for treatment of neonatal hypotension in low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 24 hours of age
* Infants with birth weight of <1001 grams and/or gestational age of <29 weeks
* Not initiated on any continuous pressor therapy prior to enrollment
* Intravenous line in place
* Outborn infants meeting eligibility criteria

Exclusion Criteria:

* Infants not meeting eligibility criteria
* Infants with life-threatening congenital defects
* Infants with congenital hydrops
* Infants with frank hypovolemia (perinatal history consistent with decreased circulating blood volume plus clinical signs of hypovolemia)
* Infants with other unresolved causes of hypotension (air leaks, lung overdistention, or metabolic abnormalities).

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle R Rios, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Rios DR, Kaiser JR. Vasopressin versus dopamine for treatment of hypotension in extremely low birth weight infants: a randomized, blinded pilot study. J Pediatr. 2015 Apr;166(4):850-5. doi: 10.1016/j.jpeds.2014.12.027. Epub 2015 Jan 29. PMID 25641242

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Started | 10 | 10 | 50
Completed | 10 | 10 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm | Total
Number analyzed (Participants) | 10 | 10 | 50 | 70
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age of subjects in weeks
  weeks | 25.1 (1) | 25.7 (2) | 25.6 (1) | 25.6 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 28 | 37
  Male | 5 | 6 | 22 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Each Group Who Have Achieved an Optimal Mean Blood Pressure Value at 24 Hours of Life
Description: Optimal mean blood pressure (OMBP) will be defined as either a 10% increase in mean blood pressure value or a 2-3 mmHg rise in mean blood pressure value AND an improvement in tissue perfusion as demonstrated by a resolution in the specified clinical symptom (designated upon enrollment) within 4-6 hours of having reached OMBP
Time Frame: 24 hours of life
Population: This outcome is only reportable in the two treatment groups as it evaluates the response to treatment of hypotension in those who received study drug. The comparison group infants were not hypotensive within the 24 hours and did not receive study drug, therefore, they are omitted from this outcome measure.
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment
Number analyzed (Participants) | 10 | 10
participants | 9 | 9

2. Secondary Outcome: Heart Rate Change From Baseline
Description: Heart rate change from baseline during study drug administration
Time Frame: 96 hours or until hypotension completely resolved and medications stopped
Population: This outcome is only reportable in the two treatment groups as it evaluates the change in heart rate in those who received study drug. The comparison group infants were not hypotensive within the 24 hours and did not receive study drug, therefore, they are omitted from this outcome measure.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Dopamine Treatment | Vasopressin Treatment
Number analyzed (Participants) | 10 | 10
beats per minute | 31 (19) | 0 (10)

3. Secondary Outcome: Acid-base Status
Time Frame: 96 hours or until hypotension resolved and medication completely stopped
Population: Treatment groups during study drug administration. Comparison group during first 96 hours of life. For all- only arterial gases
Measure: Mean (Standard Deviation); unit: pH
Groups:
- Comparison Group: Infants not diagnosed with hypotension in first 24 hours
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Group
Number analyzed (Participants) | 10 | 10 | 50
pH | 7.18 (.07) | 7.2 (.07) | 7.25 (.09)

4. Secondary Outcome: Hyponatremia
Time Frame: 96 hours or until medication completely stopped
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 3 | 3 | 11

5. Secondary Outcome: Urine Output
Time Frame: 96 hours or until hypotension resolved and medication completely stopped
Measure: Mean (Standard Deviation); unit: ml/kg/hr
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
ml/kg/hr | 4.4 (1.4) | 3.5 (1.4) | 3.9 (1.4)

6. Secondary Outcome: Evidence of Ischemic Changes
Description: Physical examinations were done on at least a twice daily basis to evaluate for any ischemic lesions (especially on the limbs) of all subjects. The presence of any lesion considered to be due to ischemia would have been reported in this data.
Time Frame: 96 hours or until medication completely stopped
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 0 | 0 | 0

7. Secondary Outcome: Necrotizing Enterocolitis
Time Frame: until hospital discharge, up to 12 weeks
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 0 | 1 | 2

8. Secondary Outcome: Ventilator Days
Time Frame: Until hospital discharge, up to 15 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
days | 52 [37 to 160] | 45.5 [23.5 to 56] | 17.5 [1 to 38]

9. Secondary Outcome: Presence of Patent Ductus Arteriosus (PDA)
Time Frame: until hospital discharge, up to 12 weeks
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 5 | 6 | 34

10. Secondary Outcome: Grade 3 Intraventricular Hemorrhage or Worse on Head Ultrasound
Time Frame: Until hospital discharge, up to 15 months
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 3 | 3 | 6

11. Secondary Outcome: Retinopathy of Prematurity Stage 3 or Higher
Description: All subjects were followed by an ophthalmologist with initial exam at 4-6 weeks of age. The Stages describe the ophthalmoscopic findings at the junction between the vascularized and avascular retina. Each subject is followed until cleared by ophthalmology. For this outcome measure, the most severe stage of disease was used in analysis.
  Stage 1 is a faint demarcation line. Stage 2 is an elevated ridge. Stage 3 is extraretinal fibrovascular proliferation (neovascularization). Stage 4 is sub-total retinal detachment. Stage 5 is total retinal detachment. Stages 1 and 2 do not lead to blindness. However, they can progress to the more severe stages.
Time Frame: Until hospital discharge, up to 15 months
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 3 | 2 | 4

12. Secondary Outcome: Presence of Bronchopulmonary Dysplasia (BPD)
Description: Infants were evaluated for oxygen need at 36 weeks postmenstrual age. If they required supplemental oxygen, they were diagnosed with BPD
Time Frame: 36 weeks postmenstrual age
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 8 | 4 | 31

13. Secondary Outcome: All Cause Mortality
Time Frame: admission to hospital discharge, up to 15 months
Measure: Number; unit: participants
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
Number analyzed (Participants) | 10 | 10 | 50
participants | 2 | 4 | 10

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, up to 15 months
Arm/Group | Dopamine Treatment | Vasopressin Treatment | Comparison Arm
All-Cause Mortality (participants affected / at risk) | 2/10 | 4/10 | 10/50
Serious Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 22/50
Other Adverse Events (participants affected / at risk) | 3/10 | 4/10 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dopamine Treatment (N=10) | Vasopressin Treatment (N=10) | Comparison Arm (N=50)
Necrotizing Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 7
Bowel Perforation (Gastrointestinal disorders) | 3 | 2 | 4
Sepsis (Infections and infestations) | 4 | 5 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dopamine Treatment (N=10) | Vasopressin Treatment (N=10) | Comparison Arm (N=50)
Hyponatremia (Renal and urinary disorders) | 3 | 4 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes